CLINICAL TRIAL: NCT01942915
Title: Safety and Efficacy Investigation of Patients With Liver Cirrhosis by Transplantation of Umbilical Cord Blood Mononuclear Cells
Brief Title: Umbilical Cord Blood Mononuclear Cells Therapy in Liver Cirrhosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Quanhai Li, Director of Cell Thearpy Center, the First Hospital of HeibeiMU, Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12276102D-Liver Cirrhosis
Record Dates: First submitted 2013-09-06; First posted 2013-09-16 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- umbilical cord blood mononuclear cells (Experimental): Umbilical Cord blood come from healthy puerpera. Erythrocyte in umbilical cord blood was separated and deleted through sedimentation. Mononuclear cells in umbilical cord blood were then isolated with a conventional method and reagent,Ficoll,by density gradient centrifugation.
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cells

INTERVENTIONS:
Biological: Umbilical Cord Blood Mononuclear Cells — Participants will be transplanted with umbilical cord blood mononuclear cells.

SUMMARY:
This study is to evaluate the safety and efficacy of umbilical cord blood mononuclear cells transplantation in liver cirrhosis patients.

DETAILED DESCRIPTION:
Decompensated liver cirrhosis (LC), a life-threatening complication of chronic liver disease, is one of the major indications for liver transplantation. Recently, umbilical cord blood mononuclear cells transfusion has been shown to lead to the regression of liver fibrosis in animal model. The investigators thus investigated the safety of the therapy with life signs like temperature, pulse, blood pressure, the incidence of hepatocellular carcinoma and mortality and so on. And the efficacy was evaluated with the measurement of alanine aminotransferase (ALT), glutamic oxaloacetic transaminase (AST), total bilirubin (TBIL), direct bilirubin (DBIL), albumin (ALB), cholinesterase (CHE), prothrombin time (PT) and child-pugh score.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hepatocirrhosis: according to the standard of child- pugh, liver functions to achieve class A or B patients, Including C class patients but can achieve B class after treatment

Exclusion Criteria:

1. Patients with C class by child-pugh score
2. Patients in the acute phase of severe hepatitis
3. Patients have been diagnosed with cancer of the liver
4. Patients with severe cardiopulmonary cerebral disease, and in the failure state
5. Patients in Highly allergic constitution
6. Patients with moderately severe mental disease

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
child-pugh classification | whinin 7 days before transplantation, 1,3 and 6 months after transplantation
  1. child-pugh A (child-pugh score 5-6)
  2. child-pugh B (child-pugh score 7-9)
  3. child-pugh C (child-pugh score≥10)

SECONDARY OUTCOMES:
coagulation | whinin 7 days before transplantation, 1,3,6 months after transplantation
  1. prothrombin time (PT)
  2. activated partial thromboplastin time (APTT)
  3. fibrinogen (FIB)
liver function | whinin 7 days before transplantation, 1,3 and 6 months after transplantation
  1. alanine aminotransferase (ALT)
  2. aspartate aminotransferase (AST)
  3. total bilirubin （TBIL）
  4. direct bilirubin (DBIL)
  5. serum cholinesterase (CHE)
  6. albumin (ALB)
vital signs | 1, 2 and 3 days after transplantation
  1. temperature
  2. pulse
  3. blood pressure
incidence of hepatocellular carcinoma | 1, 3 and 6 months after transplantation
mortality | 1, 3 and 6 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Baoyong Yan, doctor, Study Chair — The First Hospital of Hebei Medical University; Lixin Tong, master, Study Director — The First Hospital of Hebei Medical University; Sui Zhang, master, Principal Investigator — The First Hospital of Hebei Medical University; Quanhai Li, doctor, Principal Investigator — The First Hospital of Hebei Medical University
Locations (1):
- the First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China